CLINICAL TRIAL: NCT06382220
Title: Low Dose Bupivacaine Versus Prilocaine Regarding Hemodynamic Stability and Safety in Geriatrics: A Randomized, Double-Blind Comparative Study
Brief Title: Low Dose Bupivacaine Versus Prilocaine Regarding Hemodynamic Stability and Safety in Geriatrics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R550
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Recruitment
MeSH Terms: interventions — Bupivacaine; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) Bupivacaine group (Active Comparator): who received 7.5 mg (low dose) hyperbaric bupivacaine 0.5%
  Interventions: Drug: Bupivacain
- Group (B) Prilocaine group (Active Comparator): patients received 40 mg (low dose) intrathecal hyperbaric prilocaine
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — drug injection
  Other Names: prilocaine

SUMMARY:
Orthopedic interventions under spinal anesthesia is considered a common practice in elderly patients undergo surgery, and may be associated with lower risks of death, delirium,and major medical complications .

Spinal anesthesia can cause disastrous hemodynamical changes in the form of hypotension and bradycardia in elderly patients due to limited physiological reserve and presence of systemic illness . The degree of hypotension is proportional to the extent of sympathetic blockade. thus unilateral Spinal anesthesia described by Tanasichuk et AL. was used aiming to minimize these hymodynamical changes compared to bilateral block by restricting the extent of sympathetic blockade.

Bupivacaine has been used in spinal anaesthesia in orthodecic surgeries . It provides a short motor block onset time with a long motor block duration . If bupivacaine is used, the main disadvantage is the significant inter-individual variability with clinically significant differences in onset time, dermatomal spread and motor block duration . Prilocaine is a local anaesthetic agent that belongs to the same family as bupivacaine. In the last decade and with the development of day surgery, prilocaine 2% has become more commonly used for orthopaedic surgical procedures . Prilocaine induces a shorter motor block with less urinary retention, which better facilitates enhanced recovery after surgery . Usually, doses administered in spinal anaesthesia vary from 20 to 80 mg . Given the intermediate motor block duration,

The aim of this study

To compare between Unilateral low dose spinal anesthesia using bupivacaine versus prilocaine regarding hemodynamical stability and safety in below knee orthopedic surgeries in elderly people.

DETAILED DESCRIPTION:
This study will be performed in the in the FAYOUM University hospital after the local Institutional Ethics Committee and local institutional review board approval. The study design will be double-blind randomized controlled study . A detailed informed consent will be signed by the eligible patients before recruitment and randomization.

Population of Study

* Group 1 : Group (A) Bupivacaine group n = 50 patients who received 7.5 mg (low dose) hyperbaric bupivacaine 0.5% (Marcaine®, AstraZeneca, Sweden) in 2 mL volume (1.5 mL hyperbaric bupivacaine 0.5% diluted with 0.5 mL sterile distilled water) intrathecal at level lumbar L3-L4 or L4-L5 in lateral decubitus position keeping the operated side dependent and remained in this position for 10 min before turning supine.
* Group 2 : Group (B) Prilocaine group n = 50 patients received 40 mg (low dose) intrathecal hyperbaric prilocaine 2% (Takipril, Sunny Medical group, Egypt under liscense from Sintetica, Switzerland)in 2 mL volume as described in group A. The injection will be in the midline over 30 s by 25 gauge (G) Quincke needle under strict aseptic condition.

Inclusion Criteria :

100 elderly patients (60 years old or above), of either gender, with American Society of Anesthesiologists (ASA) physical status I, II, and III who were scheduled for elective knee and below knee orthopedic surgeries expected to the last for 40-60 min under spinal anesthesia.

Exclusion Criteria :

Patients height < 1.55 or > 1.75 m, with other neurological diseases, spine abnormalities, absolute, and relative contraindications to spinal anesthesia as patients suffering from intracranial hypertension, major bleeding disorder, patients on anticoagulant, local infection, dementia, and allergic reaction to local anesthetics.

Sample Size ( number of participants included ) 100 patients

Methodology in details :

All patients received Ringer's lactate infusion 5 mL/ kg and maintained intraoperatively with a rate of 5 mL/kg/h. before performance of subarachnoid blockade. Baseline heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and oxygen saturation (SpO2) were recorded. Patients were allocated to either study groups using a randomized central computer generated sequence and a sealed envelope assignment held by an investigator not involved with the clinical management or data collection, and they were randomly allocated into two groups as follows: Group (A) Bupivacaine group n = 50 patients who received 7.5 mg (low dose) hyperbaric bupivacaine 0.5% (Marcaine®, AstraZeneca, Sweden) in 2 mL volume (1.5 mL hyperbaric bupivacaine 0.5% diluted with 0.5 mL sterile distilled water) intrathecal at level lumbar L3-L4 or L4-L5 in lateral decubitus position keeping the operated side dependent and remained in this position for 10 min before turning supine. Moreover, Group (B) Prilocaine group n = 50 patients received 40 mg (low dose) intrathecal hyperbaric prilocaine 2% (Takipril, Sunny Medical group, Egypt under liscense from Sintetica, Switzerland)in 2 mL volume as described in group A. The injection will be in the midline over 30 s by 25 gauge (G) Quincke needle under strict aseptic condition. The study solution was prepared by another investigator and its content blinded to the anesthetist who administered it, the anesthesiologist who will collect the data will be unaware about any of the experimental groups. If adequate surgical anesthesia was not achieved, general anesthesia was performed, and patient was excluded from our study. HR, SBP, DBP, MAP and SpO2 were recorded every 5-minute interval until the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (60 years old or above)
* either gender
* American Society of Anesthesiologists (ASA) physical status I, II, and III who were scheduled for elective knee and below knee orthopedic surgeries expected to the last for 40-60 min under spinal anesthesia.

Exclusion Criteria:

* Patients height < 1.55 or > 1.75 m,
* with other neurological diseases, spine abnormalities,
* absolute, and relative contraindications to spinal anesthesia as patients suffering from intracranial hypertension, major bleeding disorder, patients on anticoagulant, local infection, dementia, and allergic reaction to local anesthetics.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
The rate of occurrence of hypotension | intraoperative
  mean arterial blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
NO SHARE

REFERENCES:
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Result] Neuman MD, Fleisher LA, Even-Shoshan O, Mi L, Silber JH. Nonoperative care for hip fracture in the elderly: the influence of race, income, and comorbidities. Med Care. 2010 Apr;48(4):314-20. doi: 10.1097/mlr.0b013e3181ca4126. PMID 20355262